CLINICAL TRIAL: NCT03433339
Title: Spinal Cord Stimulation for the Treatment of Major Depressive Disorder
Acronym: SPIDEP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Lindner Center of HOPE (Other); Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Francisco Romo-Nava, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIDEP 2017-7424
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder
Keywords: depression; transcutaneous spinal direct current stimulation; non-invasive; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: 8-week, double blinded, randomized, sham controlled, parallel group, pilot clinical trial study design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent operator (trained personnel from the research team) will prepare the tsDCS device parameters for each session, but will not participate in the rest of the assessments. Patients and raters will remain blinded to spinal stimulation protocol assigned to each participant throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Treatment (Experimental): Thoracic anodal transcutaneous spinal direct current stimulation 2.5 milliampere (mA) for 20 min/ three times per week for 8 weeks.
  Interventions: Device: Active transcutaneous spinal direct current stimulation
- Sham Treatment (Sham Comparator): Thoracic anodal transcutaneous spinal direct current sham stimulation session of 20min/ three times per week for 8 weeks.
  Interventions: Device: Sham transcutaneous spinal direct current stimulation

INTERVENTIONS:
Device: Active transcutaneous spinal direct current stimulation — Active anode electrodes placed at Thoracic 10 level, Cathode electrode placed on right shoulder.
  Arms: Active Treatment
Device: Sham transcutaneous spinal direct current stimulation — Sham anode electrodes placed at Thoracic 10 level, Cathode electrode placed on right shoulder.
  Arms: Sham Treatment

SUMMARY:
This pilot clinical trial will evaluate the efficacy and safety of transcutaneous direct current stimulation (tsDCS) in major depressive disorder.

DETAILED DESCRIPTION:
This study aims to 1) determine the efficacy and safety of tsDCS in adult patients with major depressive disorder (MDD) and 2) investigate interoceptive awareness, somatic symptoms, autonomic and metabolic regulation as potential mediators of antidepressant response to tsDCS. We predict that 1) Active tsDCS treatment will result in a greater decrease in depressive symptom severity compared to Sham tsDCS in adult patients with MDD, 2) active tsDCS will be safe and well tolerated in adult patients with MDD and 3) change in interoceptive awareness, somatic symptoms, and autonomic and metabolic parameters will be associated with change in depressive symptom severity. To accomplish these aims, we will conduct an 8-week, double blinded, randomized, sham controlled, parallel group, pilot clinical trial study design. A total of 20 adult antidepressant-free MDD patients will be randomized to receive Active (n=10) or Sham (n=10) tsDCS protocols for 8 weeks in a 1:1 ratio. We will combine the use of a tsDCS device, psychometric instruments to diagnose MDD, and measures of depressive symptom severity, somatic symptoms, interoceptive awareness, autonomic function (blood pressure, heart rate), and potential metabolic markers as predictors of response.

ELIGIBILITY:
Inclusion criteria:

1. age 18-55 yrs., inclusive
2. female or male
3. Body mass index (BMI) 18.5 to 35 kg/mts2, inclusive
4. current MDD episode diagnoses confirmed by Mini International Neuropsychiatric Interview (MINI) 5.0 with a duration of ≥1 month and ≤24 months
5. moderate MDD symptoms according to Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 20 to ≤35
6. no current or recent (past month) antidepressant pharmacological treatment
7. Generalized anxiety disorder (GAD) and other anxiety symptoms will be permitted
8. using an effective contraceptive method (all participants of childbearing potential).

Exclusion criteria:

1. Current or lifetime MDD episode non-responsive to two or more antidepressant treatments at adequate doses and time (including ECT)
2. Current or lifetime bipolar disorder or schizophrenia diagnosis
3. current (past month): PTSD, psychotic or substance use disorder (nicotine and caffeine allowed)
4. significant risk of suicide according to Columbia Suicide Severity Rating Scale (CSSRS) or clinical judgment, or suicidal behavior in the past year
5. current chronic severe pain conditions
6. current chronic use of: opioids analgesics, medications that affect blood pressure or drugs with significant autonomic effects (stimulants and antipsychotics allowed if dose stable for 1 month)
7. neurological, endocrinological, cardiovascular (including diagnosed hypertension) or other clinically significant medical conditions as judged by the clinician
8. skin lesions on electrode placement region
9. implanted electrical medical devices
10. Pregnancy
11. suspected Intellectual quotient (IQ)<80
12. any other clinically relevant reason as judged by the clinician.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Romo-Nava, MD,PhD, Principal Investigator — University of Cincinnati/ Lindner Center of HOPE
Locations (1):
- Lindner Center of HOPE/University of Cincinnati, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
A plan for individual participant data is not included in the current protocol. Following Federal, State and Institutional regulations, data could be shared with other researchers after the study ends.

REFERENCES:
- [Derived] Romo-Nava F, Awosika OO, Basu I, Blom TJ, Welge J, Datta A, Guillen A, Guerdjikova AI, Fleck DE, Georgiev G, Mori N, Patino LR, DelBello MP, McNamara RK, Buijs RM, Frye MA, McElroy SL. Effect of non-invasive spinal cord stimulation in unmedicated adults with major depressive disorder: a pilot randomized controlled trial and induced current flow pattern. Mol Psychiatry. 2024 Mar;29(3):580-589. doi: 10.1038/s41380-023-02349-9. Epub 2023 Dec 20. PMID 38123726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All study procedures involving participants were conducted at the Lindner Center of HOPE (affiliated with the University of Cincinnati) in Mason, Ohio, with a recruitment period from August 29, 2018, to September 13, 2022.
Pre-assignment Details: Pre-screened 671 participants. Forty two were assessed for eligibility on site. A total of 22 were excluded for not meeting eligibility criteria (n=19) or declined to participate (n=3). A total of 20 participants were randomized.
Period: Overall Study
Arm/Group | Active Treatment | Sham Treatment
Started | 10 | 10
Completed | 8 | 6
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Coronavirus disease (COVID-19) Pandemic Related Restrictions | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Although 10 participants were randomized on each arm, one participant on the Sham group withdrew after only completing the baseline visit and was excluded from the analysis. Baseline and longitudinal results analyze 10 participants on the active group and 9 on the sham group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Sham Treatment | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (9.8) | 36.8 (13.1) | 34.2 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
Montgomery Asberg Depression Rating Scale (MADRS) Score [Mean (Standard Deviation); unit: summed total scores] — Montgomery Asberg Depression Rating Scale (MADRS) score at baseline. Scores range between 0 to 60. Higher scores indicate a worse severity of symptoms.
  summed total scores | 29.0 (2.3) | 29.4 (3.8) | 29.2 (3.05)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Score Change
Description: Difference in change from baseline to week 8 (or last available observation) in Montgomery Asberg Depression Rating Scale summed total scores scores between active and sham transcutaneous spinal direct current stimulation (tsDCS) groups. Scores range from 0 to 60, with higher scores indicating worse depressive symptom severity.
Time Frame: 8 weeks (or last available observation).
Population: All participants with at least one post baseline Montgomery Asberg Depression Rating Scale total scores assessment were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: summed total scores
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
summed total scores | -21.7 (2.3) | -14.6 (2.5)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.040, ANOVA — p-value threshold for statistical significance <0.05; Mixed ANOVA model considering all available data

2. Secondary Outcome: Number of Participants With Skin Redness
Description: Number of participants with skin redness in the active and sham tsDCS groups.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment: Thoracic anodal transcutaneous spinal direct current stimulation 2.5mA for 20 min/ three times per week for 8 weeks.
  Active transcutaneous spinal direct current stimulation: Active anode electrodes placed at Thoracic 10 level, Cathode electrode placed on right shoulder.
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
Participants | 9 | 4

3. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: Clinical Global Impression-Improvement (CGI-I) scale score at week 8 (or last available information) difference between Active and Sham tsDCS groups. Range is from 1 to 7 with lower scores indicating better outcome.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: total score of the scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
total score of the scale | 1.3 (0.3) | 2.0 (0.3)

4. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Sub-component Score (Item 2) Change
Description: MADRS Item 2 score change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. MADRS Item 2 (Reported sadness) scores range from 0 to 6 and a higher score indicates a worse severity.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
score on a scale | -3.2 (0.4) | -1.8 (0.4)

5. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) Score Change
Description: PHQ-9 score change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Scores range from 0 to 27, with higher scores indicating worse severity.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
score on a scale | -12.6 (2.2) | -10.3 (2.4)

6. Secondary Outcome: Multidimensional Assessment of Interoceptive Awareness (MAIA) Score Change-Noticing Subscale
Description: MAIA Noticing subscale score change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Noticing Subscale scores range 0 to 5 and higher scores indicate better outcomes.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
score on a scale | -0.0 (0.5) | -0.2 (0.5)

7. Secondary Outcome: Binge Eating Scale (BES) Score Change
Description: BES score change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Scores range from 0 to 46, with higher scores indicating a worse outcome.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
score on a scale | -7.3 (2.7) | -3.0 (3.0)

8. Secondary Outcome: Four-Dimensional Symptom Questionnaire (4-DSQ)- Somatization Dimension Score Change
Description: 4-DSQ Somatization dimension score change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Somatization scale scores range from 0 to 32, with higher scores indicating a worse outcome.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
score on a scale | -3.3 (2.1) | -6.9 (2.3)

9. Secondary Outcome: Systolic Blood Pressure Score Change
Description: Systolic Blood Pressure score change in mmHg from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Normal range is considered below 140 mmHg. A greater decrease from baseline to week 8 in mmHg is considered favorable.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
mmHg | -5.0 (3.9) | -2.9 (4.2)

10. Secondary Outcome: Heart Rate Score Change
Description: Heart Rate score change in beats per minute (BPM) from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Normal BPM is considered between 60 to 100. A decrease in value is considered favorable.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
Beats per minute | 4.7 (3.9) | 5.3 (4.2)

11. Secondary Outcome: Body Mass Index Change
Description: Body mass index (BMI) change in kg/mts2 from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Normal range is 18 to 25 kg/mt2. A decrease in value is considered favorable.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
kg/m^2 | -0.3 (2.0) | 1.5 (2.2)

12. Secondary Outcome: Adiponectin Level Change
Description: Adiponectin level change (in ug/mL) from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. No normative levels available. Decreased levels are considered favorable in the context of the study.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: ug/mL
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
ug/mL | -805 (1640) | 1472 (2409)

13. Secondary Outcome: Leptin Level Change
Description: Leptin level (in ng/ml) change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Usual normal range 4.7 - 23.7 ng/ML. Decreased levels are considered favorable.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
ng/mL | -1.5 (4.4) | 2.7 (6.4)

14. Secondary Outcome: Cortisol Level Change
Description: Cortisol level change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Typical afternoon levels may range 5-10 nmol/L. Decreased levels are considered favorable outcomes.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
nmol/L | -0.7 (2.2) | -0.9 (3.1)

15. Secondary Outcome: Insulin Level Change
Description: Insulin level change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Fasting range typically 16-166 Milli-international Units Per Liter (mIU/L). Decreased levels are considered a favorable outcome.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Milli-international Units/ Liter (mIU/L)
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
Milli-international Units/ Liter (mIU/L) | -4.2 (4.6) | -7.2 (6.8)

16. Secondary Outcome: Fibroblast Growth Factor-21 (FGF-21) Level Change
Description: Fibroblast growth factor-21 (FGF-21) level change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Levels in ng/ml. No normative range established. Decreased levels are considered favorable in the context of the study.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
ng/ml | -13.3 (53.2) | -30.9 (78.1)

17. Secondary Outcome: Fatty Acid (LCn-3) Level Change
Description: Fatty Acid (LCn-3) level percentage change from baseline to week 8 (or last available observation) difference between Active and Sham tsDCS groups. Results reported on Erythrocyte eicosapentaenoic acid + docosahexaenoic acid (EPA+DHA) percentage change. Increase in EPA+DHA would indicate a better outcome.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 10 | 9
Percentage change | -0.02 (0.19) | -0.01 (0.22)

ADVERSE EVENTS:
Time Frame: During the eight week study duration.
Arm/Group | Active Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=10) | Sham Treatment (N=9)
Anxiety/Panic symptoms (Nervous system disorders) | 1 (1) | 1 (1)
Asymptomatic decrease in heart rate (Cardiac disorders) | 1 (1) | 0 (0)
Itching/Burnign sensation (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Cold-like symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
External Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Friction Blister in Feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Prickling Sensation (Nervous system disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin redness (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4) — Electrode site, transient.
Vaginities (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This is a proof of concept pilot feasibility clinical trial with a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT03433339/Prot_SAP_001.pdf